CLINICAL TRIAL: NCT00628199
Title: Derivation of Primary Donor Cell Lines for Human Cell Reprogramming
Brief Title: Study to Create Potential Cell-Based Therapies to Treat Human Disease and Disability
Status: Enrolling by invitation | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Marius Wernig, Professor of Pathology, Stanford University
Other Study IDs: SU-12202007-950; NCT00553826; NCT00553826 (obsolete NCT alias)
Record Dates: First submitted 2008-02-22; First posted 2008-03-04 (Estimated); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Metabolic Diseases; Infertility
MeSH Terms: conditions — Metabolic Diseases; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin sample taken from under the arm, or left over material from surgery; cells are grown out to fibroblasts then frozen

INTERVENTIONS:
Procedure: Improving the scientific process of human cell reprogramming

SUMMARY:
This is a research study in which your cells will be used for somatic cell nuclear transfer (SCNT), and/or genetic reprogramming research which may result in the production of stem cell lines. This study does not provide treatment.

DETAILED DESCRIPTION:
It is thought that studies of genetic reprogramming and SCNT using human cells have the potential to give us new basic knowledge about human development. Current work will focus on developing this basic knowledge. In the future, human embryonic stem cell lines (hESC) derived from genetic reprogramming and SCNT may also have the potential to develop into cell types that are useful for cell-based therapies to treat human disease and disability.

ELIGIBILITY:
Inclusion Criteria:1. Donors with a degenerative disease phenotype or genetic disorders such as Type I Diabetes, heart disease, or infertility (azoospermia and premature ovarian failure)

Exclusion Criteria:1. Unable to read or understand English. 2. Unable to provide skin biopsy sample due to skin condition in the underarm area.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with specific disease or infertility with potential for stem cell therapy
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-09 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marius Wernig, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States